CLINICAL TRIAL: NCT02037165
Title: Effectiveness of Two Different Doses of BI 1026706 on the Overall Peak-to-Peak (PtP) N2/P2-component Amplitude of Laser (Somatosensory, Radiant-heat) Evoked Potentials (LEP) in UVB (Ultraviolet)-Irradiated Skin in Healthy Male Volunteers (a Single-blinded, Randomised, Placebo-controlled, Single-dose, Five-way Crossover Study)
Brief Title: Effectiveness of Two Different Doses of BI 1026706 on the Overall Peak-to-Peak (PtP) N2/P2-component Amplitude of Laser (Somatosensory, Radiant-heat) Evoked Potentials (LEP) in UVB(Ultraviolet)-Irradiated Skin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1320.3; 2012-005691-33 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Pregabalin; Celecoxib

ARMS (5):
- Test Treatment 1: BI 1026706 (Experimental): BI 1026706 plus matching placebo to BI 1026706 Powder for Oral Solution (PfOS) and placebo tablet
  Interventions: Drug: Placebo to BI 1026706; Drug: BI 1026706
- Test Treatment 2: BI 1026706 (Experimental): BI 1026706 and placebo tablet
  Interventions: Drug: Placebo to BI 1026706; Drug: BI 1026706
- Reference Treatment 1: BI 1026706 (Experimental): Matching placebo to BI 1026706 PfOS and placebo tablet
  Interventions: Drug: Placebo to BI 1026706
- Reference Treatment 2: Celecoxib (Experimental): Celecoxib hard capsule as active comparator plus matching placebo to BI 1026706 PfOS
  Interventions: Drug: Placebo to BI 1026706; Drug: Celecoxib
- Reference Treatment 3: Pregabalin (Experimental): Pregabalin hard capsule as active comparator plus matching placebo to BI 1026706 PfOS
  Interventions: Drug: Placebo to BI 1026706; Drug: Pregabalin

INTERVENTIONS:
Drug: Placebo to BI 1026706 — Placebo tablet
Drug: Pregabalin — Pregabalin hard capsule
  Arms: Reference Treatment 3: Pregabalin
Drug: BI 1026706 — BI 1026706 oral solution
  Arms: Test Treatment 1: BI 1026706; Test Treatment 2: BI 1026706
Drug: Celecoxib — Celecoxib hard capsule
  Arms: Reference Treatment 2: Celecoxib

SUMMARY:
* To investigate the influence of different doses of BI 1026706 on the primary endpoint (PtP-amplitude LEP in UV skin) compared to placebo.
* The comparison of both doses of BI 1026706 to celecoxib in the UVB treatment.
* Comparison of both doses of BI 1026706 to placebo and pregabalin in the capsaicin treatment
* Exploration of the pharmacokinetics of BI 1026706
* Exploration of safety and tolerability of BI 1026706

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the investigator's assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (Blood Pressure, Pulse Rate), 12-lead electrocardiogram, and clinical laboratory
2. Age 18 to 55 years (incl.)
3. BMI (Body Mass Index) 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

1. Any finding in the medical examination (including Blood Pressure, Pulse Rate or Electrocardiogram) deviating from normal and judged clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug(s)
7. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2014-04-09 (Actual); Study Completion 2014-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1320.3.1 Boehringer Ingelheim Investigational Site, Dörnach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg: Single dose administration per treatment. A washout period of at least 6 days was required between the treatments. Treatment sequence A: 50mg BI 1026706 (powder for oral solution [PfOS]), 200mg BI 1026706 (PfOS), placebo (matching placebo to BI 1026706), 200mg Celecoxib (Cele, hard capsule), 150mg Pregabalin (Preg, hard capsule). Mode of admin.: oral with 200 mL of water.
- 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo: Single dose administration per treatment. A washout period of at least 6 days was required between the treatments. Treatment sequence B: 200mg BI 1026706 (PfOS), 50mg BI 1026706 (PfOS), 200mg Cele (hard capsule), 150mg Preg (hard capsule), placebo (matching placebo).Mode of admin.: oral with 200 mL of water.
- Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele: Single dose administration per treatment. A washout period of at least 6 days was required between the treatments. Treatment sequence C: placebo (matching placebo), 150mg Preg (hard capsule), 50mg BI 1026706 (PfOS), 200mg BI 1026706 (PfOS), 200mg Cele (hard capsule). Mode of admin.: oral with 200 mL of water.
- 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706: Single dose administration per treatment. A washout period of at least 6 days was required between the treatments. Treatment sequence D: 200mg Cele (hard capsule), placebo (matching placebo), 150mg Preg (hard capsule), 50mg BI 1026706 (PfOS), 200mg BI 1026706 (PfOS). Mode of admin.: oral with 200 mL of water.
- 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706: Single dose administration per treatment. A washout period of at least 6 days was required between the treatments. Treatment sequence E: 150mg Preg (hard capsule), 200mg Cele (hard capsule), 200mg BI 1026706 (PfOS), placebo (matching placebo), 50mg BI 1026706 (PfOS). Mode of admin.: oral with 200 mL of water.
Period: Period 1 (2 Days)
Arm/Group | 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706
Started | 5 (randomized subjects) | 5 (randomized subjects) | 5 (randomized subjects) | 5 (randomized subjects) | 5 (randomized subjects)
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (6 Days)
Arm/Group | 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2 (2 Days)
Arm/Group | 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (6 Days)
Arm/Group | 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3 (2 Days)
Arm/Group | 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 (6 Days)
Arm/Group | 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4 (2 Days)
Arm/Group | 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout Period 4 (6 Days)
Arm/Group | 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Period: Period 5 (2 Days)
Arm/Group | 50mg BI1026706/200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706
Started | 5 | 5 | 5 | 5 | 4
Completed | 5 | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) : all subjects who were dispensed study medication and were documented to have taken at least 1 dose of study drug.
Groups:
- 50mg BI1026706/ 200mg BI1026706/Placebo/200mg Cele/150mg Preg: Single dose administration per treatment. A washout period of at least 6 days was required between the treatments. Treatment sequence A: 50mg BI 1026706 (PfOS), 200mg BI 1026706 (PfOS), placebo (matching placebo to BI 1026706), 200mg Celecoxib (Cele, hard capsule), 150mg Pregabalin (Preg, hard capsule). Mode of admin.: oral with 200 mL of water.
- 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo: Single dose administration per treatment. A washout period of at least 6 days was required between the treatments. Treatment sequence B: 200mg BI 1026706 (PfOS), 50mg BI 1026706 (PfOS), 200mg Cele (hard capsule), 150mg Preg (hard capsule), placebo (matching placebo). Mode of admin.: oral with 200 mL of water.
- 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706: Single dose administration per treatment. A washout period of at least 6 days was required between the treatments. Treatment sequence E: 150mg Preg (hard capsule), 200mg Cele (hard capsule), 200mg BI 1026706 (hard capsule), placebo (matching placebo), 50mg BI 1026706 (PfOS). Mode of admin.: oral with 200 mL of water.
- Total: Total of all reporting groups
Arm/Group | 50mg BI1026706/ 200mg BI1026706/Placebo/200mg Cele/150mg Preg | 200mg BI1026706/50mg BI1026706/200mg Cele/150mg Preg/Placebo | Placebo/150mg Preg/50mg BI1026706/200mg BI1026706/200mg Cele | 200mg Cele/Placebo/150mg Preg/50mg BI1026706/200mg BI1026706 | 150mg Preg/200mg Cele/200mg BI1026706/Placebo/50mg BI1026706 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (10.3) | 35.8 (11.6) | 41.2 (10.9) | 35.0 (11.2) | 32.8 (7.9) | 35.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 5 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Peak-to-Peak(PtP) N2/P2-component Amplitude of Laser (Somatosensory/Radiant Heat) Evoked Potentials (LEP) in Ultraviolet B (UVB) -Irradiated Skin
Description: Overall Peak-to-Peak (PtP) N2/P2-component amplitude of Laser (somatosensory/radiant heat) evoked potentials (LEP) in UVB-irradiated skin.
  Treated set (TS)
Time Frame: up to 24 hours (h): -2:05h, 0:30h, 1:00h, 2:00h, 3:00h, 4:00h, 5:00h, 6:00h, 22:00h, 24:00h (relative to study drug administration [h:min])
Population: pharmacodynamic set(PDS): included all subjects from the TS who provided in any treatment period a baseline value and at least 1 PD profile post drug administration for the primary or secondary PD endpoint, which was considered evaluable, and without (important) protocol violation(s) with respect to the statistical evaluation of PD endpoints.
Measure: Mean (Standard Deviation); unit: Microvolts (µv)
Groups:
- Placebo: Matching placebo to BI 1026706, Mode of Administration: Oral with 200 mL of water.
- 50 mg BI 1026706: treatment group: 50 mg BI 1026706, powder for oral solution (PfOS), Mode of Admin.: Oral with 200 mL of water.
- 200 mg BI 1026706: treatment group: 200 mg BI 1026706, powder for oral solution (PfOS), Mode of Admin.: Oral with 200 mL of water.
- 200 mg Celecoxib (Cele): 200 mg Celecoxib (cele), hard capsule, single dose, mode of admin.: oral with 200 mL of water.
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 200 mg Celecoxib (Cele)
Number analyzed (Participants) | 25 | 24 | 25 | 25
Microvolts (µv)
  at -2:05h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at -2:05h | 29.22 (8.98) | 26.08 (10.41) | 28.93 (8.06) | 26.35 (9.22)
  at 0:30h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 0:30h | 27.84 (8.83) | 28.00 (10.67) | 24.88 (8.69) | 26.60 (8.90)
  at 1:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 1:00h | 25.57 (10.02) | 27.11 (8.64) | 26.77 (10.31) | 27.60 (9.31)
  at 2:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 2:00h | 26.74 (8.51) | 28.78 (8.81) | 29.03 (9.04) | 24.87 (7.11)
  at 3:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 3:00h | 29.48 (9.50) | 30.93 (7.39) | 29.02 (7.98) | 25.05 (8.32)
  at 4:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 4:00h | 30.54 (8.77) | 31.40 (10.90) | 31.44 (8.42) | 23.97 (7.71)
  at 5:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 5:00h | 31.74 (10.07) | 30.10 (8.37) | 30.79 (9.84) | 24.10 (8.78)
  at 6:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 6:00h | 32.16 (10.48) | 28.12 (8.29) | 29.04 (10.66) | 26.77 (8.61)
  at 22:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 22:00h | 34.48 (10.97) | 32.51 (8.30) | 34.50 (10.97) | 33.06 (11.33)
  at 24:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 24:00h | 34.43 (16.61) | 32.83 (9.62) | 32.98 (12.31) | 30.03 (10.54)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BI 1026706; A repeated measures model was applied to the change from baseline of the endpoint which included the fixed effects 'period', 'treatment', 'mean of the period baselines of primary PD endpoint', 'baseline of primary PD endpoint of the respective period', and 'session', the random effect 'subject', and the interaction terms 'mean of the period baselines × session', 'baseline of the respective period × session', 'period × session', and 'treatment × session'; Test type: Superiority or Other; adjusted mean difference = 1.12, 95% CI 2-sided [-3.0 to 5.2], Standard Error of Mean 2.0801 — Adjusted mean treatment difference between 50 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 0:30h after the dose administration
Statistical Analysis 2: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 2.66, 95% CI 2-sided [-1.4 to 6.8], Standard Error of Mean 2.0796 — Adjusted mean treatment difference between 50 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 1:00h after the dose administration
Statistical Analysis 3: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 3.00, 95% CI 2-sided [-1.1 to 7.1], Standard Error of Mean 2.0792 — Adjusted mean treatment difference between 50 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 2:00h after the dose administration
Statistical Analysis 4: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 2.53, 95% CI 2-sided [-1.6 to 6.6], Standard Error of Mean 2.0790 — Adjusted mean treatment difference between 50 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 3:00h after the dose administration
Statistical Analysis 5: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.72, 95% CI 2-sided [-2.4 to 5.8], Standard Error of Mean 2.0789 — Adjusted mean treatment difference between 50 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 4:00h after the dose administration
Statistical Analysis 6: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.15, 95% CI 2-sided [-4.2 to 3.9], Standard Error of Mean 2.0790 — Adjusted mean treatment difference between 50 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 5:00h after the dose administration
Statistical Analysis 7: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -3.15, 95% CI 2-sided [-7.2 to 0.9], Standard Error of Mean 2.0792 — Adjusted mean treatment difference between 50 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 6:00h after the dose administration
Statistical Analysis 8: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.31, 95% CI 2-sided [-5.4 to 2.8], Standard Error of Mean 2.0796 — Adjusted mean treatment difference between 50 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 22:00h after the dose administration
Statistical Analysis 9: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.15, 95% CI 2-sided [-4.2 to 3.9], Standard Error of Mean 2.0801 — Adjusted mean treatment difference between 50 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 24:00h after the dose administration
Statistical Analysis 10: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -2.68, 95% CI 2-sided [-6.7 to 1.3], Standard Error of Mean 2.0282 — Adjusted mean treatment difference between 200 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 0:30h after the dose administration
Statistical Analysis 11: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.58, 95% CI 2-sided [-2.4 to 5.6], Standard Error of Mean 2.0279 — Adjusted mean treatment difference between 200 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 1:00h after the dose administration
Statistical Analysis 12: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 2.63, 95% CI 2-sided [-1.4 to 6.6], Standard Error of Mean 2.0278 — Adjusted mean treatment difference between 200 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 2:00h after the dose administration
Statistical Analysis 13: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.17, 95% CI 2-sided [-4.2 to 3.8], Standard Error of Mean 2.0277 — Adjusted mean treatment difference between 200 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 3:00h after the dose administration
Statistical Analysis 14: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.20, 95% CI 2-sided [-2.8 to 5.2], Standard Error of Mean 2.0276 — Adjusted mean treatment difference between 200 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 4:00h after the dose administration
Statistical Analysis 15: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.59, 95% CI 2-sided [-4.6 to 3.4], Standard Error of Mean 2.0277 — Adjusted mean treatment difference between 200 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 5:00h after the dose administration
Statistical Analysis 16: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -2.88, 95% CI 2-sided [-6.9 to 1.1], Standard Error of Mean 2.0278 — Adjusted mean treatment difference between 200 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 6:00h after the dose administration
Statistical Analysis 17: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.43, 95% CI 2-sided [-3.6 to 4.4], Standard Error of Mean 2.0279 — Adjusted mean treatment difference between 200 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 22:00h after the dose administration
Statistical Analysis 18: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.04, 95% CI 2-sided [-5.0 to 2.9], Standard Error of Mean 2.0282 — Adjusted mean treatment difference between 200 mg BI 1026706 and placebo in the change from baseline. This analysis represents the results evaluated at 24:00h after the dose administration

2. Secondary Outcome: Overall Peak-to-Peak (PtP) N2/P2-component Amplitude of (LEP) in Capsaicin-irritated Skin
Description: Overall Peak-to-Peak (PtP) N2/P2-component amplitude of (LEP) in capsaicin-irritated skin.
Time Frame: up to 24 hours(h): -1:20h, 0:30h, 1:00h, 2:00h, 3:00h, 4:00h, 5:00h, 6:00h, 22:00h, 24:00h (relative to study drug administration [h:min])
Population: PDS
Measure: Mean (Standard Deviation); unit: µv
Groups:
- 150 mg Pregabalin (Prega): 150 mg pregabalin (prega) hard capsule, single dose, mode of admin.: oral with 200 mL of water.,
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 150 mg Pregabalin (Prega)
Number analyzed (Participants) | 25 | 24 | 25 | 25
µv
  at -1:20h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at -1:20h | 21.17 (10.33) | 18.53 (6.88) | 19.57 (9.24) | 22.44 (10.94)
  at 0:30h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 0:30h | 27.21 (10.36) | 25.00 (9.69) | 25.35 (9.12) | 25.20 (10.61)
  at 1:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 1:00h | 27.96 (9.38) | 23.67 (10.49) | 23.11 (8.96) | 24.80 (9.89)
  at 2:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 2:00h | 27.97 (9.32) | 23.94 (8.40) | 24.98 (7.29) | 24.83 (10.89)
  at 3:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 3:00h | 27.69 (8.74) | 25.68 (8.20) | 26.13 (9.35) | 24.46 (9.58)
  at 4:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 4:00h | 27.53 (9.19) | 26.74 (6.99) | 25.26 (8.33) | 22.76 (9.37)
  at 5:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 5:00h | 26.25 (9.39) | 25.81 (9.44) | 25.31 (8.06) | 23.00 (10.03)
  at 6:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 6:00h | 25.77 (9.10) | 24.14 (8.33) | 24.06 (8.24) | 23.30 (9.18)
  at 22:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 22:00h | 26.75 (9.00) | 24.46 (9.07) | 23.53 (8.44) | 23.15 (8.24)
  at 24:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 24:00h | 24.83 (8.77) | 22.94 (8.06) | 23.91 (11.18) | 22.59 (9.71)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.94, 95% CI 2-sided [-4.6 to 2.7], Standard Error of Mean 1.8566 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -2.87, 95% CI 2-sided [-6.5 to 0.8], Standard Error of Mean 1.8560 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -3.08, 95% CI 2-sided [-6.7 to 0.6], Standard Error of Mean 1.8557 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.63, 95% CI 2-sided [-5.3 to 2.0], Standard Error of Mean 1.8555 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.11, 95% CI 2-sided [-3.5 to 3.8], Standard Error of Mean 1.8554 — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.66, 95% CI 2-sided [-3.0 to 4.3], Standard Error of Mean 1.8555 — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.19, 95% CI 2-sided [-4.8 to 2.5], Standard Error of Mean 1.8557 — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.34, 95% CI 2-sided [-5.0 to 2.3], Standard Error of Mean 1.8560 — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.84, 95% CI 2-sided [-4.5 to 2.8], Standard Error of Mean 1.8566 — [estimate comment as in outcome 1, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.10, 95% CI 2-sided [-4.7 to 2.5], Standard Error of Mean 1.8257 — [estimate comment as in outcome 1, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -3.98, 95% CI 2-sided [-7.6 to -0.4], Standard Error of Mean 1.8254 — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -2.43, 95% CI 2-sided [-6.0 to 1.2], Standard Error of Mean 1.8252 — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.29, 95% CI 2-sided [-4.9 to 2.3], Standard Error of Mean 1.8251 — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Slope = -1.72, 95% CI 2-sided [-5.3 to 1.9], Standard Error of Mean 1.8250 — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.23, 95% CI 2-sided [-3.8 to 3.4], Standard Error of Mean 1.8251 — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 16: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.46, 95% CI 2-sided [-5.0 to 2.1], Standard Error of Mean 1.8252 — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -2.65, 95% CI 2-sided [-6.2 to 0.9], Standard Error of Mean 1.8254 — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.31, 95% CI 2-sided [-3.9 to 3.3], Standard Error of Mean 1.8257 — [estimate comment as in outcome 1, analysis 18]

3. Secondary Outcome: Single "Peripheral" N2-component Amplitudes - Measured in UVB-irradiated Skin Type
Description: Single "peripheral" N2-component amplitudes - measured in UVB-irradiated skin type.
Time Frame: up to 24 hours(h): -2:05h, 0:30h, 1:00h, 2:00h, 3:00h, 4:00h, 5:00h, 6:00h, 22:00h, 24:00h (relative to study drug administration [h:min])
Population: PDS
Measure: Mean (Standard Deviation); unit: µv
Groups:
- 200 mg Celecoxib (Cele): 200 mg celecoxib (cele) hard capsule, single dose, mode of admin.: oral with 200 mL of water.
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 200 mg Celecoxib (Cele)
Number analyzed (Participants) | 25 | 24 | 25 | 25
µv
  at -2:05h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at -2:05h | 14.62 (4.02) | 12.78 (6.42) | 14.25 (4.73) | 13.45 (5.61)
  at 0:30h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 0:30h | 14.48 (5.01) | 13.77 (6.03) | 12.70 (4.99) | 13.62 (4.55)
  at 1:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 1:00h | 12.54 (5.15) | 14.42 (5.76) | 13.45 (5.34) | 14.29 (4.67)
  at 2:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 2:00h | 14.40 (4.37) | 14.90 (5.50) | 15.06 (4.48) | 12.22 (3.59)
  at 3:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 3:00h | 16.08 (4.74) | 16.85 (5.08) | 14.58 (3.93) | 12.61 (4.36)
  at 4:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 4:00h | 16.52 (4.99) | 16.92 (5.37) | 16.95 (4.27) | 11.87 (4.35)
  at 5:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 5:00h | 17.20 (5.37) | 16.87 (4.81) | 16.93 (5.69) | 12.07 (4.68)
  at 6:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 6:00h | 17.46 (5.77) | 15.51 (5.28) | 15.30 (4.94) | 14.04 (5.51)
  at 22:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 22:00h | 18.71 (6.36) | 17.12 (5.23) | 18.93 (6.11) | 16.99 (6.35)
  at 24:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 24:00h | 19.01 (8.69) | 17.74 (5.31) | 18.58 (6.55) | 16.67 (5.84)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.16, 95% CI 2-sided [-2.8 to 2.5], Standard Error of Mean 1.3652 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 2.18, 95% CI 2-sided [-0.5 to 4.9], Standard Error of Mean 1.3652 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.01, 95% CI 2-sided [-1.7 to 3.7], Standard Error of Mean 1.3652 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.26, 95% CI 2-sided [-1.4 to 3.9], Standard Error of Mean 1.3652 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.71, 95% CI 2-sided [-2.0 to 3.4], Standard Error of Mean 1.3652 — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.36, 95% CI 2-sided [-2.3 to 3.0], Standard Error of Mean 1.3652 — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.58, 95% CI 2-sided [-4.3 to 1.1], Standard Error of Mean 1.3652 — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.51, 95% CI 2-sided [-4.2 to 1.2], Standard Error of Mean 1.3652 — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.83, 95% CI 2-sided [-3.5 to 1.8], Standard Error of Mean 1.3652 — [estimate comment as in outcome 1, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.64, 95% CI 2-sided [-4.2 to 1.0], Standard Error of Mean 1.3254 — [estimate comment as in outcome 1, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.07, 95% CI 2-sided [-1.5 to 3.7], Standard Error of Mean 1.3253 — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.82, 95% CI 2-sided [-1.8 to 3.4], Standard Error of Mean 1.3253 — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.32, 95% CI 2-sided [-3.9 to 1.3], Standard Error of Mean 1.3253 — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.56, 95% CI 2-sided [-2.0 to 3.2], Standard Error of Mean 1.3254 — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.04, 95% CI 2-sided [-2.6 to 2.6], Standard Error of Mean 1.3253 — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 16: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -2.05, 95% CI 2-sided [-4.7 to 0.6], Standard Error of Mean 1.3253 — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.40, 95% CI 2-sided [-2.2 to 3.0], Standard Error of Mean 1.3253 — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.26, 95% CI 2-sided [-2.9 to 2.3], Standard Error of Mean 1.3254 — [estimate comment as in outcome 1, analysis 18]

4. Secondary Outcome: Single "Peripheral" N2-component Amplitudes - Measured in Capsaicin-irritated Skin Type
Description: Single "peripheral" N2-component amplitudes - measured in capsaicin-irritated skin type.
Time Frame: as for outcome 2
Population: PDS
Measure: Mean (Standard Deviation); unit: µv
Groups:
- 150 mg Pregabalin (Prega): 150 mg pregabalin (prega) hard capsule, single dose, mode of admin.: oral with 200 mL of water.
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 150 mg Pregabalin (Prega)
Number analyzed (Participants) | 25 | 24 | 25 | 25
µv
  at -1:20h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at -1:20h | 10.42 (5.76) | 9.65 (4.63) | 9.27 (5.47) | 10.99 (5.89)
  at 0:30h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 0:30h | 13.95 (5.59) | 12.73 (5.03) | 12.17 (5.30) | 12.17 (6.39)
  at 1:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 1:00h | 13.70 (5.27) | 11.43 (5.83) | 11.50 (5.48) | 12.03 (5.34)
  at 2:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 2:00h | 13.77 (5.39) | 11.85 (4.94) | 12.36 (4.43) | 12.18 (6.26)
  at 3:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 3:00h | 13.44 (5.07) | 12.71 (5.59) | 13.39 (5.23) | 12.51 (6.20)
  at 4:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 4:00h | 13.52 (4.40) | 13.54 (4.58) | 12.63 (4.20) | 10.86 (6.05)
  at 5:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 5:00h | 12.93 (4.11) | 13.01 (5.65) | 12.84 (4.70) | 11.49 (6.45)
  at 6:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 6:00h | 12.36 (5.43) | 12.27 (5.52) | 12.27 (4.46) | 12.03 (5.39)
  at 22:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 22:00h | 13.59 (5.03) | 12.84 (5.68) | 11.53 (4.95) | 11.77 (5.39)
  at 24:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 24:00h | 13.18 (5.83) | 11.71 (4.87) | 11.70 (5.66) | 11.35 (5.53)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.96, 95% CI 2-sided [-3.4 to 1.5], Standard Error of Mean 1.2419 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.97, 95% CI 2-sided [-4.4 to 0.5], Standard Error of Mean 1.2418 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.64, 95% CI 2-sided [-4.1 to 0.8], Standard Error of Mean 1.2418 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.55, 95% CI 2-sided [-3.0 to 1.9], Standard Error of Mean 1.2418 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = 0.29, 95% CI 2-sided [-2.1 to 2.7], Standard Error of Mean 1.2418 — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = 0.39, 95% CI 2-sided [-2.1 to 2.8], Standard Error of Mean 1.2418 — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = 0.11, 95% CI 2-sided [-2.3 to 2.6], Standard Error of Mean 1.2418 — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.54, 95% CI 2-sided [-3.0 to 1.9], Standard Error of Mean 1.2418 — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.12, 95% CI 2-sided [-3.6 to 1.3], Standard Error of Mean 1.2419 — [estimate comment as in outcome 1, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.29, 95% CI 2-sided [-3.7 to 1.1], Standard Error of Mean 1.2344 — [estimate comment as in outcome 1, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.89, 95% CI 2-sided [-4.3 to 0.5], Standard Error of Mean 1.2343 — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.16, 95% CI 2-sided [-3.6 to 1.3], Standard Error of Mean 1.2343 — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = 0.09, 95% CI 2-sided [-2.3 to 2.5], Standard Error of Mean 1.2343 — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.72, 95% CI 2-sided [-3.1 to 1.7], Standard Error of Mean 1.2343 — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = 0.42, 95% CI 2-sided [-2.0 to 2.8], Standard Error of Mean 1.2343 — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 16: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = 0.13, 95% CI 2-sided [-2.3 to 2.6], Standard Error of Mean 1.2343 — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.71, 95% CI 2-sided [-4.1 to 0.7], Standard Error of Mean 1.2343 — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.18, 95% CI 2-sided [-3.6 to 1.2], Standard Error of Mean 1.2344 — [estimate comment as in outcome 1, analysis 18]

5. Secondary Outcome: Single "Central" P2-component Amplitudes - Measured in UVB-irradiated Skin Type
Description: Single "central" P2-component amplitudes - measured in UVB-irradiated skin type.
Time Frame: as for outcome 3
Population: PDS
Measure: Mean (Standard Deviation); unit: µv
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 200 mg Celecoxib (Cele)
Number analyzed (Participants) | 25 | 24 | 25 | 25
µv
  UVB, at -2:05h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at -2:05h | 14.59 (6.57) | 13.31 (5.43) | 14.68 (4.83) | 12.90 (5.08)
  UVB, at 0:30h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at 0:30h | 14.06 (6.24) | 14.23 (6.26) | 12.18 (4.82) | 12.98 (5.86)
  UVB, at 1:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at 1:00h | 13.03 (6.66) | 12.69 (5.21) | 13.32 (6.28) | 13.31 (5.52)
  UVB, at 2:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at 2:00h | 12.34 (5.79) | 13.88 (5.30) | 13.97 (5.99) | 12.65 (4.56)
  UVB, at 3:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at 3:00h | 13.40 (6.37) | 14.08 (4.99) | 14.44 (6.16) | 12.44 (5.59)
  UVB, at 4:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at 4:00h | 14.01 (6.07) | 14.49 (7.11) | 14.49 (6.04) | 12.10 (5.11)
  UVB, at 5:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at 5:00h | 14.54 (6.53) | 13.23 (5.38) | 13.87 (6.71) | 12.03 (5.81)
  UVB, at 6:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at 6:00h | 14.71 (6.58) | 12.61 (5.16) | 13.74 (7.30) | 12.73 (4.95)
  UVB, at 22:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at 22:00h | 15.77 (6.59) | 15.40 (5.36) | 15.57 (8.02) | 16.07 (6.61)
  UVB, at 24:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  UVB, at 24:00h | 15.43 (9.07) | 15.09 (6.23) | 14.40 (7.63) | 13.36 (5.73)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.79, 95% CI 2-sided [-1.5 to 3.1], Standard Error of Mean 1.1758 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.51, 95% CI 2-sided [-1.8 to 2.8], Standard Error of Mean 1.1755 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 2.06, 95% CI 2-sided [-0.2 to 4.4], Standard Error of Mean 0.1752 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.33, 95% CI 2-sided [-1.0 to 3.6], Standard Error of Mean 1.1751 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.12, 95% CI 2-sided [-1.2 to 3.4], Standard Error of Mean 1.1750 — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.57, 95% CI 2-sided [-2.9 to 1.7], Standard Error of Mean 1.1751 — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.43, 95% CI 2-sided [-3.7 to 0.9], Standard Error of Mean 1.1752 — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.24, 95% CI 2-sided [-2.1 to 2.5], Standard Error of Mean 1.1755 — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.43, 95% CI 2-sided [-1.9 to 2.7], Standard Error of Mean 1.1758 — [estimate comment as in outcome 1, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.68, 95% CI 2-sided [-4.0 to 0.6], Standard Error of Mean 1.1567 — [estimate comment as in outcome 1, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.52, 95% CI 2-sided [-1.8 to 2.8], Standard Error of Mean 1.1566 — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.89, 95% CI 2-sided [-0.4 to 4.2], Standard Error of Mean 1.1565 — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 1.25, 95% CI 2-sided [-1.0 to 3.5], Standard Error of Mean 1.1564 — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.67, 95% CI 2-sided [-1.6 to 2.9], Standard Error of Mean 1.1564 — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference of 200 mg BI mi = -0.43, 95% CI 2-sided [-2.7 to 1.8], Standard Error of Mean 1.1564 — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 16: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.76, 95% CI 2-sided [-3.0 to 1.5], Standard Error of Mean 1.1565 — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 0.09, 95% CI 2-sided [-2.2 to 2.4], Standard Error of Mean 1.1566 — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.71, 95% CI 2-sided [-3.0 to 1.6], Standard Error of Mean 1.1567 — [estimate comment as in outcome 1, analysis 18]

6. Secondary Outcome: Single "Central" P2-component Amplitudes - Measured in Capsaicin-irritated Skin Type
Description: Single "central" P2-component amplitudes - measured in capsaicin-irritated skin type.
Time Frame: as for outcome 2
Population: PDS
Measure: Mean (Standard Deviation); unit: µv
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 150 mg Pregabalin (Prega)
Number analyzed (Participants) | 25 | 24 | 25 | 25
µv
  at -1:20h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at -1:20h | 10.75 (5.43) | 8.88 (3.80) | 10.30 (4.51) | 11.45 (6.12)
  at 0:30h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 0:30h | 13.83 (6.53) | 12.27 (5.76) | 13.18 (5.22) | 13.03 (5.59)
  at 1:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 1:00h | 14.25 (5.64) | 12.24 (5.86) | 11.61 (4.56) | 12.77 (5.67)
  at 2:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 2:00h | 14.20 (5.41) | 12.09 (4.18) | 12.62 (4.10) | 12.65 (5.09)
  at 3:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 3:00h | 14.25 (5.24) | 12.97 (4.18) | 12.74 (5.02) | 11.94 (4.78)
  at 4:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 4:00h | 14.01 (6.07) | 13.20 (4.20) | 12.63 (4.74) | 11.90 (4.95)
  at 5:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 5:00h | 13.32 (5.89) | 12.79 (4.94) | 12.47 (4.63) | 11.51 (4.60)
  at 6:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 6:00h | 13.41 (5.07) | 11.87 (3.91) | 11.78 (4.76) | 11.27 (4.93)
  at 22:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 22:00h | 13.16 (5.03) | 11.62 (4.91) | 12.00 (5.00) | 11.38 (4.60)
  at 24:00h: number analyzed (Participants) | 24 | 24 | 25 | 25
  at 24:00h | 11.65 (3.83) | 11.24 (3.91) | 12.21 (6.54) | 11.24 (5.35)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.53, 95% CI 2-sided [-2.7 to 1.7], Standard Error of Mean 1.1242 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.99, 95% CI 2-sided [-3.2 to 1.2], Standard Error of Mean 1.1240 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.45, 95% CI 2-sided [-3.7 to 0.8], Standard Error of Mean 1.1238 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.06, 95% CI 2-sided [-3.3 to 1.2], Standard Error of Mean 1.1236 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.10, 95% CI 2-sided [-2.3 to 2.1], Standard Error of Mean 1.1236 — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.08, 95% CI 2-sided [-2.3 to 2.1], Standard Error of Mean 1.1236 — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.50, 95% CI 2-sided [-3.7 to 0.7], Standard Error of Mean 1.1238 — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.05, 95% CI 2-sided [-3.3 to 1.2], Standard Error of Mean 1.1240 — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.07, 95% CI 2-sided [-2.3 to 2.1], Standard Error of Mean 1.1242 — [estimate comment as in outcome 1, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.35, 95% CI 2-sided [-2.5 to 1.8], Standard Error of Mean 1.0986 — [estimate comment as in outcome 1, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -2.31, 95% CI 2-sided [-4.5 to -0.2], Standard Error of Mean 1.0985 — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.39, 95% CI 2-sided [-3.6 to 0.8], Standard Error of Mean 1.0984 — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.38, 95% CI 2-sided [-3.5 to 0.8], Standard Error of Mean 1.0984 — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.15, 95% CI 2-sided [-3.3 to 1.0], Standard Error of Mean 1.0983 — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.63, 95% CI 2-sided [-2.8 to 1.5], Standard Error of Mean 1.0984 — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 16: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -1.53, 95% CI 2-sided [-3.7 to 0.6], Standard Error of Mean 1.0984 — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -0.96, 95% CI 2-sided [-3.1 to 1.2], Standard Error of Mean 1.0985 — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = 0.76, 95% CI 2-sided [-1.4 to 2.9], Standard Error of Mean 1.0986 — [estimate comment as in outcome 1, analysis 18]

7. Secondary Outcome: Electronic Visual Analogue Scale (VAS) (100mm VAS "Post Laser Pain" Scales) - Measured in the UVB-irradiated Skin Type
Description: Electronic Visual Analogue Scale (100mm VAS "Post Laser Pain" scales) - measured in the UVB-irradiated skin type, where 0mm = 'no pain' and 100mm = 'severe pain'.
Time Frame: as for outcome 3
Population: PDS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 200 mg Celecoxib (Cele)
Number analyzed (Participants) | 25 | 24 | 25 | 25
units on a scale
  at -2:05h | 30.40 (16.71) | 28.42 (16.67) | 30.16 (19.01) | 35.08 (18.93)
  at 0:30h | 39.24 (18.16) | 32.46 (19.71) | 32.24 (19.60) | 38.00 (19.56)
  at 1:00h | 41.48 (17.44) | 36.67 (21.94) | 37.16 (21.40) | 38.28 (20.15)
  at 2:00h | 50.56 (22.04) | 42.92 (23.54) | 46.88 (21.44) | 44.00 (19.84)
  at 3:00h | 56.40 (23.90) | 53.25 (24.78) | 55.52 (27.33) | 52.72 (24.24)
  at 4:00h | 62.16 (22.96) | 56.33 (24.64) | 62.04 (27.73) | 56.68 (26.64)
  at 5:00h | 66.60 (25.31) | 63.71 (24.33) | 65.48 (27.90) | 56.52 (25.23)
  at 6:00h | 69.24 (23.97) | 65.46 (25.26) | 66.60 (27.20) | 56.48 (25.61)
  at 22:00h | 61.68 (24.53) | 57.13 (25.61) | 57.76 (26.54) | 59.28 (25.10)
  at 24:00h | 65.00 (24.39) | 61.96 (26.70) | 61.13 (27.51) | 61.96 (27.20)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -6.13, 95% CI 2-sided [-12.5 to 0.2], Standard Error of Mean 3.2064 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -3.88, 95% CI 2-sided [-10.6 to 2.9], Standard Error of Mean 3.4032 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -6.67, 95% CI 2-sided [-13.3 to -0.0], Standard Error of Mean 3.3393 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.80, 95% CI 2-sided [-8.9 to 5.3], Standard Error of Mean 3.5727 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -4.43, 95% CI 2-sided [-10.7 to 1.8], Standard Error of Mean 3.1554 — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.18, 95% CI 2-sided [-6.4 to 4.0], Standard Error of Mean 2.6161 — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -2.35, 95% CI 2-sided [-8.7 to 4.0], Standard Error of Mean 3.1849 — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -2.78, 95% CI 2-sided [-10.3 to 4.7], Standard Error of Mean 3.7688 — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.27, 95% CI 2-sided [-7.0 to 4.4], Standard Error of Mean 2.8570 — [estimate comment as in outcome 1, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -6.91, 95% CI 2-sided [-13.2 to -.07], Standard Error of Mean 3.1527 — [estimate comment as in outcome 1, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -4.22, 95% CI 2-sided [-10.9 to 2.4], Standard Error of Mean 3.3457 — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -3.61, 95% CI 2-sided [-10.1 to 2.9], Standard Error of Mean 3.2806 — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.80, 95% CI 2-sided [-7.8 to 6.2], Standard Error of Mean 3.5078 — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.05, 95% CI 2-sided [-6.2 to 6.1], Standard Error of Mean 3.0965 — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -1.05, 95% CI 2-sided [-6.1 to 4.0], Standard Error of Mean 2.5649 — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 16: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -2.59, 95% CI 2-sided [-8.8 to 3.7], Standard Error of Mean 3.1250 — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -3.84, 95% CI 2-sided [-11.2 to 3.5], Standard Error of Mean 3.7013 — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -3.05, 95% CI 2-sided [-8.7 to 2.6], Standard Error of Mean 2.8201 — [estimate comment as in outcome 1, analysis 18]

8. Secondary Outcome: Electronic Visual Analogue Scale (100mm VAS "Post Laser Pain" Scales) - Measured in the Capsaicin-irritated Skin Type.
Description: Electronic Visual Analogue Scale (100mm VAS "Post Laser Pain" scales) - measured in the capsaicin-irritated skin type, where 0mm = 'no pain' and 100mm = 'severe pain'.
Time Frame: as for outcome 2
Population: PDS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 150 mg Pregabalin (Prega)
Number analyzed (Participants) | 25 | 24 | 25 | 25
units on a scale
  at -1:20h | 18.64 (13.66) | 16.79 (11.69) | 20.36 (18.33) | 22.60 (16.74)
  at 0:30h | 30.64 (17.93) | 25.96 (16.73) | 27.92 (19.42) | 31.28 (18.80)
  at 1:00h | 35.48 (17.70) | 30.08 (16.68) | 33.76 (20.68) | 32.80 (19.65)
  at 2:00h | 39.52 (18.71) | 32.79 (19.76) | 36.92 (21.38) | 32.16 (17.27)
  at 3:00h | 46.44 (20.02) | 38.79 (20.03) | 44.52 (26.01) | 37.16 (18.68)
  at 4:00h | 47.48 (21.92) | 41.79 (19.14) | 48.40 (26.97) | 40.92 (20.25)
  at 5:00h | 49.16 (21.51) | 44.29 (19.78) | 47.56 (26.15) | 43.92 (21.63)
  at 6:00h | 50.48 (24.91) | 47.21 (20.84) | 47.00 (25.03) | 41.56 (20.64)
  at 22:00h | 38.52 (20.13) | 34.29 (19.67) | 39.48 (23.71) | 36.32 (18.81)
  at 24:00h | 39.92 (19.96) | 36.83 (20.12) | 38.60 (22.70) | 37.80 (18.65)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -3.78, 95% CI 2-sided [-8.9 to 1.3], Standard Error of Mean 2.5753 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -4.74, 95% CI 2-sided [-9.8 to 0.3], Standard Error of Mean 2.5162 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -6.06, 95% CI 2-sided [-11.9 to -0.3], Standard Error of Mean 2.9156 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -6.83, 95% CI 2-sided [-13.8 to 0.1], Standard Error of Mean 3.4987 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -5.24, 95% CI 2-sided [-12.6 to 2.1], Standard Error of Mean 3.6922 — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -4.71, 95% CI 2-sided [-11.9 to 2.5], Standard Error of Mean 3.6166 — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -3.09, 95% CI 2-sided [-10.5 to 4.3], Standard Error of Mean 3.7073 — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -3.82, 95% CI 2-sided [-12.1 to 4.5], Standard Error of Mean 4.1860 — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -2.67, 95% CI 2-sided [-9.5 to 4.1], Standard Error of Mean 3.4254 — [estimate comment as in outcome 1, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -3.64, 95% CI 2-sided [-8.7 to 1.4], Standard Error of Mean 2.5461 — [estimate comment as in outcome 1, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -2.46, 95% CI 2-sided [-7.4 to 2.5], Standard Error of Mean 2.4848 — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -3.27, 95% CI 2-sided [-9.0 to 2.5], Standard Error of Mean 2.8811 — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -2.91, 95% CI 2-sided [-9.8 to 4.0], Standard Error of Mean 3.4569 — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = 0.27, 95% CI 2-sided [-7.0 to 7.5], Standard Error of Mean 3.6471 — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -2.27, 95% CI 2-sided [-9.4 to 4.8], Standard Error of Mean 3.5708 — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 16: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -4.21, 95% CI 2-sided [-11.5 to 3.1], Standard Error of Mean 3.6602 — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = 0.54, 95% CI 2-sided [-7.7 to 8.8], Standard Error of Mean 4.1389 — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted mean difference = -2.04, 95% CI 2-sided [-8.8 to 4.7], Standard Error of Mean 3.3835 — [estimate comment as in outcome 1, analysis 18]

9. Secondary Outcome: Weighted Needle (Pain) Threshold (WNT) in the Secondary Flare Area of Capsaicin-irritated Skin
Description: Weighted needle (pain) threshold (WNT) in the secondary flare area of capsaicin-irritated skin. The weighted needle (pain) threshold (WNT) will be determined (with regard to investigation of mechanical hyperalgesia in the secondary hyperalgesia zone around the primary capsaicin application zone) by fixed weight steps - contact made by "rounded" needle tip to skin (ranging from 1 mN to 512 mN).
Time Frame: as for outcome 2
Population: PDS
Measure: Mean (Standard Deviation); unit: millinewton (mN)
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 150 mg Pregabalin (Prega)
Number analyzed (Participants) | 25 | 24 | 25 | 25
millinewton (mN)
  at -1:20h | 348.72 (131.75) | 366.65 (123.95) | 369.98 (142.20) | 347.12 (133.57)
  at 0:30h | 312.88 (137.29) | 295.65 (126.48) | 285.78 (122.17) | 301.48 (157.97)
  at 1:00h | 290.28 (144.08) | 285.35 (144.26) | 262.20 (117.10) | 280.38 (160.61)
  at 2:00h | 269.70 (139.49) | 287.94 (148.70) | 225.48 (112.11) | 254.70 (150.10)
  at 3:00h | 274.30 (148.21) | 265.58 (147.81) | 222.66 (119.98) | 265.51 (145.58)
  at 4:00h | 268.38 (148.57) | 265.77 (151.62) | 235.15 (114.60) | 255.45 (140.19)
  at 5:00h | 261.50 (140.44) | 270.27 (157.88) | 228.09 (122.48) | 266.83 (141.25)
  at 6:00h | 292.30 (158.11) | 281.21 (163.78) | 234.30 (124.55) | 273.42 (125.06)
  at 22:00h | 331.76 (152.45) | 313.77 (159.07) | 274.92 (125.73) | 330.26 (147.94)
  at 24:00h | 323.38 (138.05) | 312.85 (156.45) | 277.38 (148.59) | 340.76 (147.36)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -29.67, 95% CI 2-sided [-88.3 to 29.0], Standard Error of Mean 29.5691 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -16.29, 95% CI 2-sided [-75.5 to 42.9], Standard Error of Mean 29.8613 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = 7.63, 95% CI 2-sided [-42.2 to 57.5], Standard Error of Mean 25.1035 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -20.47, 95% CI 2-sided [-66.7 to 25.8], Standard Error of Mean 23.3110 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -12.63, 95% CI 2-sided [-58.6 to 33.4], Standard Error of Mean 23.1894 — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -0.67, 95% CI 2-sided [-47.8 to 46.5], Standard Error of Mean 23.7285 — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -19.27, 95% CI 2-sided [-74.3 to 35.7], Standard Error of Mean 27.6359 — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -25.23, 95% CI 2-sided [-79.9 to 29.5], Standard Error of Mean 27.5524 — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs 50 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -17.19, 95% CI 2-sided [-70.9 to 36.5], Standard Error of Mean 27.0135 — [estimate comment as in outcome 1, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -39.62, 95% CI 2-sided [-97.7 to 18.5], Standard Error of Mean 29.3023 — [estimate comment as in outcome 1, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -37.06, 95% CI 2-sided [-95.7 to 21.6], Standard Error of Mean 29.5797 — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -52.45, 95% CI 2-sided [-101.8 to -3.1], Standard Error of Mean 24.8429 — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -59.87, 95% CI 2-sided [-105.6 to -14.1], Standard Error of Mean 23.0541 — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -39.96, 95% CI 2-sided [-85.5 to 5.5], Standard Error of Mean 22.9336 — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -38.99, 95% CI 2-sided [-85.6 to 7.6], Standard Error of Mean 23.4683 — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 16: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -63.69, 95% CI 2-sided [-118.1 to -9.3], Standard Error of Mean 27.3484 — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -61.36, 95% CI 2-sided [-115.6 to -7.2], Standard Error of Mean 27.2866 — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs 200 mg BI 1026706; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; adjusted mean difference = -49.40, 95% CI 2-sided [-102.6 to 3.8], Standard Error of Mean 26.7541 — [estimate comment as in outcome 1, analysis 18]

ADVERSE EVENTS:
Time Frame: From the start day of trial medication administration to Day 3 ( 3 days after the last trial medication)
Groups:
- 50 mg BI 1026706: treatment group: 50 mg BI 1026706
- 200 mg BI 1026706: treatment group: 200 BI 1026706
- 200 mg Celecoxib: treatment group: 200 mg celecoxib
- 150 mg Pregabalin: treatment group: 150 mg pregabalin
Arm/Group | Placebo | 50 mg BI 1026706 | 200 mg BI 1026706 | 200 mg Celecoxib | 150 mg Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/25 | 2/24 | 3/25 | 2/25 | 17/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | 50 mg BI 1026706 (N=24) | 200 mg BI 1026706 (N=25) | 200 mg Celecoxib (N=25) | 150 mg Pregabalin (N=25)
Sinus bradycardia (Cardiac disorders) | 3 | 2 | 3 | 2 | 5
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 8
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 9
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.